CLINICAL TRIAL: NCT01562327
Title: A Multi-national, Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab Actemra
Brief Title: A Non-interventional Study of RoActemra/Actemra (Tocilizumab) in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28142
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tocilizumab: Participants with moderate to severe rheumatoid arthritis (RA) received Tocilizumab according to individualized physician-prescribed regimens.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants received tocilizumab according to individualized physician-prescribed regimens.
  Other Names: Actemra

SUMMARY:
This multi-center, observational study will evaluate the clinical practice patterns, efficacy and safety of RoActemra/Actemra (tocilizumab) in participants with moderate to severe rheumatoid arthritis. Data will be collected from each eligible participant initiated on RoActemra/Actemra treatment by their treating physician according to local label for 6 months from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Moderate to severe rheumatoid arthritis
* Participants initiating treatment with RoActemra/Actemra on their physician's decision (in accordance with the local label), including participants who started treatment with RoActemra/Actemra in the 8 weeks prior to the enrolment visit

Exclusion Criteria:

* RoActemra/Actemra treatment more than 8 weeks prior to the enrolment visit
* Previous RoActemra/Actemra treatment in a clinical trial or for compassionate use
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis participants treated with tocilizumab
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Argentina (6):
  - Buenos Aires
  - Ciudad Autonoma de
  - La Plata
  - San Juan
  - San Juan Bautista
  - San Miguel de Tucumán

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab
Started | 50
Completed | 42
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Participant drop-out | 1
Not completed — Infusion not received at 6 month window | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Tocilizumab Treatment at 6 Months After Treatment Initiation
Time Frame: 6 months after treatment initiation
Population: The Full Analysis Set (FAS) was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tocilizumab: Participants with moderate to severe RA received Tocilizumab according to individualized physician-prescribed regimens.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants | 84 [71 to 93]

2. Secondary Outcome: Percentage of Participants With Systemic Manifestations of RA at Baseline
Description: Systemic manifestations of RA included anemia, fatigue, conventional risk factors for cardiovascular disease, C-Reactive Protein (CRP) above upper limit of normal, rheumatoid nodules, rheumatoid vasculitis and interstitial lung disease. Participants were included if they experienced at least one of the conditions.
Time Frame: Baseline
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants | 40

3. Secondary Outcome: Number of Participants Who Stopped Disease-Modifying Antirheumatic Drugs (DMARDs) Prior to Start of Tocilizumab
Time Frame: Baseline
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
participants | 5

4. Secondary Outcome: Percentage of Participants Who Previously Received DMARDs
Time Frame: Baseline
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants
  0 DMARDs | 48.00
  1 DMARD | 24.00
  2 DMARDs | 14.00
  3 DMARDs | 10.00
  4 DMARDs | 0.00
  5 DMARDs | 1
  6 DMARDs | 2.00
  7 DMARDs | 0.00
  8 DMARDs | 0.00
  9 DMARDs | 0.00
  10 DMARDs | 0.00
  11 DMARDs | 2.00

5. Secondary Outcome: Reason for DMARDs Withdrawal at Baseline
Time Frame: Baseline
Population: FAS defined as all participants who received at least one dose of Tocilizumab. Number of participants analyzed signifies the participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 5
participants
  Adverse event | 2
  Unknown | 2
  Other - reason not specified | 1

6. Secondary Outcome: Number of Participants Who Stopped Biologic Agents Prior to Start of Tocilizumab
Time Frame: Baseline
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
participants | 19

7. Secondary Outcome: Percentage of Participants Who Previously Received Biologic Agents
Time Frame: Baseline
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants
  0 Biologic Agents | 62.00
  1 Biologic Agent | 16.00
  2 Biologic Agents | 16.00
  3 Biologic Agents | 4.00
  4 Biologic Agents | 2.00

8. Secondary Outcome: Reason for Biologic Agent Withdrawal at Baseline
Time Frame: Baseline
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 19
participants
  Lack of efficacy | 13
  Adverse event | 1
  Other - reason not specified | 2
  Unknown | 3

9. Secondary Outcome: Reasons for Dose Modifications
Time Frame: approximately 3 years
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
participants
  Adverse Event | 1
  Other | 21

10. Secondary Outcome: Percentage of Participants Who Discontinued From Tocilizumab for Safety Versus Efficacy
Time Frame: Approximately 3 years
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants
  Adverse Event | 4
  Lack of Efficacy | 2

11. Secondary Outcome: Percentage of Participants on Tocilizumab as Monotherapy or Combination Therapy
Description: Percentage of participants on Tocilizumab as monotherapy or combination therapy (with DMARDs) were reported at start of treatment and at 6 months from the start of treatment.
Time Frame: Baseline, Month 6
Population: FAS was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants
  Monotherapy at baseline | 14
  With DMARDs at baseline | 86
  Monotherapy at Month 6 | 14
  With DMARDs at Month 6 | 86

12. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Month 3 and Month 6
Description: The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1, for 28 joints and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 28. A decrease in score indicated improvement.
Time Frame: Baseline, Month 3, Month 6
Population: FAS was defined as all participants who received at least one dose of Tocilizumab. Here, 'n' represents the number of participants with a measure at the specified time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 29
units on a scale
  Baseline (n=29) | 12 [2 to 28]
  Change at Month 3 (n=22) | -6 [-25 to 4]
  Change at Month 6 (n=22) | -9 [-22 to 4]

13. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Month 3 and Month 6
Description: The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1, for 28 joints and were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 28. A decrease in score indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 12
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 29
units on a scale
  Baseline (n=29) | 8 [1 to 17]
  Change at Month 3 (n=22) | -5 [-16 to 4]
  Change at Month 6 (n=22) | -7.50 [-17 to 6]

14. Secondary Outcome: Disease Activity Score-28 (DAS 28) Response Classification at Month 3 and Moth 6
Description: DAS28 was calculated from SJC and TJC using 28 joints count, erythrocyte sedimentation rate (ESR) (millimeter per hour [mm/hr]), and patient global assessment of disease activity (PGH) (measured on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS) where 0=no disease activity and 100=worst disease activity). DAS28 is a measurement of RA activity on a 0 to 10 scale: a score greater than (>) 5.1 indicates high disease activity; a score between 3.2 and 5.1 indicates moderate disease activity; a score of less than 3.2 indicates low disease activity; a score of less than (<) 2.6 is considered remission.
Time Frame: Month 3, Month 6
Population: FAS was defined as all participants who received at least one dose of Tocilizumab. Number of participants analyzed signifies the participants who were evaluable for this outcome measure. Here, 'n' represents the number of participants with a measure at the specified time point.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 4
participants
  < 2.6 Clinical Remission at Month 3 (n=2) | 0
  <2.6 Clinical Remission at Month 6 (n=4) | 0
  >=2.6-<=3.2 Low Disease Activity at Month 3 (n=2) | 0
  >=2.6-<=3.2 Low Disease Activity at Month 6 (n=4) | 3
  >3.2-<=5.1 Moderate Disease at Month 3(n=2) | 2
  >3.2-<=5.1 Moderate Disease at Month 6 (n=4) | 1
  >5.1 High Disease Activity at Month 3 (n=2) | 0
  >5.1 High Disease Activity at Month 6 (n=4) | 0

15. Secondary Outcome: Clinical Disease Activity Index (CDAI) Response Classification at Month 3 and Month 6
Description: CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and physician global assessment of disease activity (PhGH) assessed on 0-10 cm VAS; 0 = no disease activity and 10 = worst disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: Month 3, Month 6
Population: FAS was defined as all participants who received at least one dose of Tocilizumab. Number of participants analyzed signifies the participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
participants
  <= 2.8 Clinical remission at Month 3 | 1
  <= 2.8 Clinical remission at Month 6 | 2
  > 2.8 and <= 10.0 Low disease activity at Month 3 | 7
  > 2.8 and <= 10.0 Low disease activity at Month 6 | 7
  > 10.0 and <= 22.0 Moderate activity at Month 3 | 6
  > 10.0 and <= 22.0 Moderate activity at Month 6 | 9
  > 22.0 High disease activity at Month 3 | 9
  > 22.0 High disease activity at Month 6 | 5

16. Secondary Outcome: Simplified Disease Activity (SDAI) Response Classification
Description: The SDAI was a combined index for measuring disease activity in RA which reflected the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and PhGH, assessed on 0-100 mm VAS where 0 = no disease activity and 100 = worst disease activity, and C-reactive protein (CRP). SDAI total score = 0-86. A SDAI score </= 3.3 represented clinical remission, a score of between 3.4 and 11.0 represented low disease activity, a score between 11 and 26.0 represented moderate disease activity and a score > 26.0 represented high (or severe) disease.
Time Frame: Month 3, Month 6
Population: Data was not collected, hence not reported.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

17. Secondary Outcome: European League Against Rheumatism (EULAR) Response
Description: Clinical response assessed as per EULAR categorical DAS28 response criteria was defined as clinically meaningful improvement at a particular time point. EULAR response was based on change from baseline (CFB) in the DAS28 score and also on the actual DAS28 score at the time point so was more reflective of the current status of the participant. The DAS28 score was a measure of the participant's disease activity, based on the TJC (28 joints), SJC (28 joints), PGH, and ESR. DAS28 total scores ranged from 0 to approximately 10. Scores <2.6 = best disease control and scores >5.1 = worse disease control. A negative CFB indicated clinically meaningful improvement. EULAR Good response: DAS28 <=3.2 and a CFB <-1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a CFB < -0.6 to ≥ -1.2. EULAR No response: DAS28 ≤3.2 or CFB greater than or equal to (>=) -0.6, DAS28 >3.2 to <=5.1 or CFB>=-0.6 and DAS28 >5.1 or CFB >=-0.6.
Time Frame: Month 3, Month 6
Population: Data was not collected, hence not reported.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

18. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) Response at Month 3 and Month 6
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR20 response required at least a 20% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: patient's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), Acute phase reactant (CRP or ESR). A reduction in the level of and acute phase reactants was considered an improvement. ACR50, ACR70, ACR90 require a 50%, 70%, 90% improvement from baseline respectively.
Time Frame: Month 3, Month 6
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 22
percentage of participants
  ACR 20 at Month 3 (n=21) | 38.10
  ACR 20 at Month 6 (n=22) | 68.18
  ACR 50 at Month 3 (n=21) | 23.81
  ACR 50 at Month 6 (n=22) | 40.91
  ACR 70 at Month 3 (n=21) | 14.29
  ACR 70 at Month 6 (n=22) | 13.64
  ACR 90 at Month 3 (n=21) | 0.00
  ACR 90 at Month 6 (n=22) | 9.09

19. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Month 3 and Month 6
Description: The physician's global assessment of disease activity was assessed using a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Month 3, Month 6
Population: FAS was defined as all participants who received at least one dose of Tocilizumab. Here, 'n' represents the number of participants with a measurement at the specified time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 35
units on a scale
  Baseline (n=35) | 51 [5 to 90]
  Change at Month 3 (n=29) | -10 [-85 to 31]
  Change at Month 6 (n=27) | -20 [-87 to 0]

20. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Month 3 and Month 6
Description: The Patient Global Assessment of disease activity provides an overall assessment of how RA affects the participant using a visual analogue score, where 0 indicates they are managing very well and 100 indicates they are managing very poorly. A decrease in the score indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 39
units on a scale
  Baseline (n=39) | 65 [5 to 100]
  Change at Month 3 (n=31) | -10 [-85 to 40]
  Change at Month 6 (n=30) | -15 [-86 to 20]

21. Secondary Outcome: Percentage of Participants With Clinical Remission in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI was a participant self-reported questionnaire for assessing the extent of a participant's functional ability. It consisted of 20 questions in 8 categories (dressing and grooming, rising, eating, walking, reach, grip, hygiene, and carrying out daily activities). Each question had 4 response options, ranging from 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. The HAQ-DI scale was an average of all the scores and ranged from 0 to 3, where higher scores represented higher disease activity.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 33
percentage of participants
  < 0.5 Clinical Remission at Baseline (n=33) | 6.06
  >= 0.5 No remission at Baseline (n=33) | 93.94
  < 0.5 Clinical Remission at Month 3 (n=25) | 40.00
  >= 0.5 No remission at Month 3 (n=25) | 60.00
  < 0.5 Clinical Remission at Month 6 (n=26) | 26.92
  >= 0.5 No remission at Month 6 (n=26) | 73.08

22. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Fatigue at Month 3 and Month 6
Description: The Patient Global Assessment of fatigue provides an overall assessment of the level of fatigue that the participant is experiencing using a visual analogue score, where 0 indicates no fatigue and 100 indicates extreme fatigue. A decrease in the score indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 28
units on a scale
  Baseline (n=28) | 70 [0 to 100]
  Change at Month 3 (n=23) | -35 [-100 to 38]
  Change at Month 6 (n=22) | -30 [-90 to 70]

23. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Pain at Month 3 and Month 6
Description: The Patient Global Assessment of pain provides an overall assessment of the severity of pain that the participant is experiencing using a visual analogue score, where 0 indicates no pain and 100 indicates unbearable pain. A decrease in the score indicates improvement.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 37
units on a scale
  Baseline (n=37) | 80 [15 to 100]
  Change at Month 3 (n=30) | -23 [-100 to 27]
  Change at Month 6 (n=29) | -25 [-95 to 24]

24. Secondary Outcome: Change From Baseline in Patient's Severity of Morning Stiffness at Month 3 and Month 6
Description: Morning stiffness was defined by the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was as limber as he/she would be during a day involving typical activities. Morning stiffness was assessed on a 100 mm VAS, where 0= none and 100= very severe.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 19
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 21
units on a scale
  Baseline (n=21) | 60 [0 to 100]
  Change at Month 3 (n=16) | -50 [-100 to 60]
  Change at Month 6 (n=14) | -25 [-87 to 10]

25. Secondary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study drug.
Time Frame: approximately 3 years
Population: Safety population was defined as all participants who received at least one dose of Tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants | 56.00

ADVERSE EVENTS:
Time Frame: Approximately 3 years
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study drug.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=50)
Femur fracture (Injury, poisoning and procedural complications) | 1
Angina unstable (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.